CLINICAL TRIAL: NCT03706560
Title: Professional Consequences of Ocular Trauma Hospitalized at the University Hospital Centre of Clermont-Ferrand
Brief Title: Professional Consequences of Ocular Trauma Hospitalized at the Hospital Centre of Clermont-Ferrand
Acronym: HOT-WORK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-399; 2018-A00605-50 (Other: 2018-A00605-50)
Record Dates: First submitted 2018-07-05; First posted 2018-10-16 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Eye Injuries; Work Performance; Occupational Stress
Keywords: workers; eye injuries; work abilities
MeSH Terms: conditions — Eye Injuries; Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ocular trauma are a real public health issue. According to WHO, it is estimates at 750,000 hospital admissions per year in the world for ocular trauma, including 200,000 for open globe injuries in the world. Consequences can be severe with a significant number of definitive low vision or blindness which can lead to professionnal reclassifications for active patients. However, no study exists on professional consequences of those ocular trauma. Some studies showed that fonctionnal loss of an eye can also have psychological consequences such as post traumatic depression or can impair the quality of life but studies are scarce on this subject.

The primary objective is to study the professional reclassification of workers at least 6 months after their hospitalization for ocular trauma.

Secondary objectives are to assess, at least 6 months after an hospitalized ocular trauma, characteristics of eye injuries, characteristics of patients, mid-term consequences at work after eye injury and on personal aspects.

DETAILED DESCRIPTION:
Use of the ophthalmologic consultation report, the ophthalmologic hospitalization report and a telephone questionnaire to carry out the study.

At least 6 months after the traumatism, an ophthalmologist member of the team, M. Vincent Jawad, will call each patient for answering a telephone questionnaire after obtention of his oral consent.

If the traumatism occur after the beginning of the study, the patient will be informed, by M. Vincent Jawad, of the modalities of the study during his hospitalization and an information letter will be given to the patient in the same time (annex 2). His non opposition will be asked by telephone, remote from the hospitalization, before proceeding to the telephone questionnaire.

If the traumatism occur before the beginning of the study or if the information and non opposition letter has not been given to the patient during the hospitalization, the information letter (annex 2) will be sent by mail to the patient before the telephone call.

In all cases, the patient's consent (or non opposition) will be collected orally before proceeding to the telephone questionnaire (annex 1).

Medical data will be obtained from the medical report of hospitalization and the last report consultation of his ophthalmologist.

ELIGIBILITY:
Inclusion Criteria:

* Adults, with a job
* hospitalized for ocular trauma in the ophthalmology unit of the University Hospital of Clermont-ferrand
* from january the first of 2005 to december the 31st of 2022.

Exclusion Criteria:

* Patient without job at the time of the ocular traumatism
* Refusal to participate in the study
* Unable to answer to the telephone questionnaire (difficulties understanding, cognitive disorders…)
* Impossibility to contact the patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, with a job, hospitalized for ocular trauma in the ophthalmology unit of the University Hospital of Clermont-ferrand from january the first of 2005 to december the 31st of 2022.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Professionnal status of workers after the ocular trauma telephone questionnaire) | at 6 months
  The professional status of workers at least 6 months after the ocular trauma, at the period of realization of the telephone questionnaire by questioning the patient; qualitative scale: reinstatement in the same workstation, adaptation of the workstation, change of work (in the same company or in an other one), no return to work.

SECONDARY OUTCOMES:
Far final visual acuity | at 6 months
  Far final visual acuity with Monoyer scale (telephone questionnaire) (in decimal).
Mecanism of ocular trauma | at least 6 months after their hospitalization for ocular trauma
  traumatism by foreign body, percussion, burn, fall, other
Initial ocular lesions | at day 1
  corneal wound, scleral wound, cataract, wounds of the lid margin, of the lacrymal ducts, hyphaema, ocular hypertension, intravitreal haemorrhage, ulceration, others
Final ocular sequelae | at 6 month
  All ocular complications that may have an impact on the final visual fonction (qualitative scale)
Proportion of work-related ocular trauma | at 6 month
  Proportion of work-related ocular trauma
Wear of protective eyewear during traumatism | at 6 month
  Wear of protective eyewear during traumatism, binary scale (yes/no)
Medical opinion of professional aptitude made by the occupational physician during work resumption examination | at 6 month
  Qualitative scale (apt, unfit with professional reclassification, dismissal for professional inability with formal contraindication of job retention)
Total duration of Work stoppage | at 6 month
  days
Variations of time of work since the ocular trauma | at 6 month
  hours per week
State of Stress and Mood at work, before and after the ocular trauma, by graduating scales (telephone questionnaire) | at 6 month
  by graduating scales, between 0 to 10, before and after the ocular trauma
Quality of sleep, before and after the ocular trauma by graduating scales (telephone questionnaire) | at 6 month
  by graduating scales, between 0 to 10, before and after the ocular trauma
Job demand, job control and social support (derived from the Karasek questionnaire) | at 6 month
  by graduating scales, between 0 to 10, before and after the ocular trauma (telephone questionnaire)
Tobacco consumption | at 6 month
  number of cigarette per day, before and after the ocular trauma
Alcohol consumption | at 6 month
  before and after the ocular trauma, in number of alcohol unity per day
Consumption of pharmaceuticals | at 6 month
  type of pharmaceuticals and any modification before and after the ocular trauma
Limitations or modifications on sport | at 6 month
  by graduated scales (between 0 to 4) (telephone questionnaire)
Limitations or modifications on driving | at 6 month
  by graduated scales (between 0 to 4) (telephone questionnaire)
Limitations or modifications on hobbies | at 6 month
  by graduated scales (between 0 to 4) (telephone questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DUTHEIL, MD,PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Negrel AD, Thylefors B. The global impact of eye injuries. Ophthalmic Epidemiol. 1998 Sep;5(3):143-69. doi: 10.1076/opep.5.3.143.8364. PMID 9805347
- [Background] Xiang H, Stallones L, Chen G, Smith GA. Work-related eye injuries treated in hospital emergency departments in the US. Am J Ind Med. 2005 Jul;48(1):57-62. doi: 10.1002/ajim.20179. PMID 15940717
- [Background] Pizzarello LD. Ocular trauma: time for action. Ophthalmic Epidemiol. 1998 Sep;5(3):115-6. doi: 10.1076/opep.5.3.115.8366. No abstract available. PMID 9805344
- [Background] Pinna A, Atzeni G, Patteri P, Salvo M, Zanetti F, Carta F. Epidemiology, visual outcome, and hospitalization costs of open globe injury in northern Sardinia, Italy. Ophthalmic Epidemiol. 2007 Sep-Oct;14(5):299-305. doi: 10.1080/09286580701198753. PMID 17994439
- [Background] Byhr E. Perforating eye injuries in a western part of Sweden. Acta Ophthalmol (Copenh). 1994 Feb;72(1):91-7. doi: 10.1111/j.1755-3768.1994.tb02744.x. PMID 8017204
- [Background] Schrader WF. [Epidemiology of open globe eye injuries: analysis of 1026 cases in 18 years]. Klin Monbl Augenheilkd. 2004 Aug;221(8):629-35. doi: 10.1055/s-2004-813254. German. PMID 15343446
- [Background] Casson RJ, Walker JC, Newland HS. Four-year review of open eye injuries at the Royal Adelaide Hospital. Clin Exp Ophthalmol. 2002 Feb;30(1):15-8. doi: 10.1046/j.1442-9071.2002.00484.x. PMID 11885788
- [Background] Tielsch JM, Parver L, Shankar B. Time trends in the incidence of hospitalized ocular trauma. Arch Ophthalmol. 1989 Apr;107(4):519-23. doi: 10.1001/archopht.1989.01070010533025. PMID 2705918
- [Background] Parver LM, Dannenberg AL, Blacklow B, Fowler CJ, Brechner RJ, Tielsch JM. Characteristics and causes of penetrating eye injuries reported to the National Eye Trauma System Registry, 1985-91. Public Health Rep. 1993 Sep-Oct;108(5):625-32. PMID 8210260
- [Background] Thylefors B. Epidemiological patterns of ocular trauma. Aust N Z J Ophthalmol. 1992 May;20(2):95-8. doi: 10.1111/j.1442-9071.1992.tb00718.x. PMID 1389141
- [Background] Cillino S, Casuccio A, Di Pace F, Pillitteri F, Cillino G. A five-year retrospective study of the epidemiological characteristics and visual outcomes of patients hospitalized for ocular trauma in a Mediterranean area. BMC Ophthalmol. 2008 Apr 22;8:6. doi: 10.1186/1471-2415-8-6. PMID 18430231
- [Background] Forrest KY, Cali JM. Epidemiology of lifetime work-related eye injuries in the U.S. population associated with one or more lost days of work. Ophthalmic Epidemiol. 2009 May-Jun;16(3):156-62. doi: 10.1080/09286580902738175. PMID 19437310
- [Background] Baillif S, Paoli V. [Open-globe injuries and intraocular foreign bodies involving the posterior segment]. J Fr Ophtalmol. 2012 Feb;35(2):136-45. doi: 10.1016/j.jfo.2011.08.003. Epub 2012 Jan 9. French. PMID 22226765
- [Background] Yuksel H, Turkcu FM, Ahin M, Cinar Y, Cingu AK, Ozkurt Z, Bez Y, Caca H. Vision-related quality of life in patients after ocular penetrating injuries. Arq Bras Oftalmol. 2014 Apr;77(2):95-8. doi: 10.5935/0004-2749.20140024. PMID 25076473
- [Background] Alexander DA, Kemp RV, Klein S, Forrester JV. Psychiatric sequelae and psychosocial adjustment following ocular trauma: a retrospective pilot study. Br J Ophthalmol. 2001 May;85(5):560-2. doi: 10.1136/bjo.85.5.560. PMID 11316717
- [Background] Schrader WF. Open globe injuries: epidemiological study of two eye clinics in Germany, 1981-1999. Croat Med J. 2004 Jun;45(3):268-74. PMID 15185415
- [Background] Rofail M, Lee GA, O'Rourke P. Quality of life after open-globe injury. Ophthalmology. 2006 Jun;113(6):1057.e1-3. doi: 10.1016/j.ophtha.2006.02.042. No abstract available. PMID 16751044
- [Background] Chandola T, Britton A, Brunner E, Hemingway H, Malik M, Kumari M, Badrick E, Kivimaki M, Marmot M. Work stress and coronary heart disease: what are the mechanisms? Eur Heart J. 2008 Mar;29(5):640-8. doi: 10.1093/eurheartj/ehm584. Epub 2008 Jan 23. PMID 18216031
- [Background] Chikani V, Reding D, Gunderson P, McCarty CA. Psychosocial work characteristics predict cardiovascular disease risk factors and health functioning in rural women: the Wisconsin Rural Women's Health Study. J Rural Health. 2005 Fall;21(4):295-302. doi: 10.1111/j.1748-0361.2005.tb00098.x. PMID 16294651
- [Background] Collins SM, Karasek RA, Costas K. Job strain and autonomic indices of cardiovascular disease risk. Am J Ind Med. 2005 Sep;48(3):182-93. doi: 10.1002/ajim.20204. PMID 16094616
- [Background] de Jonge J, Bosma H, Peter R, Siegrist J. Job strain, effort-reward imbalance and employee well-being: a large-scale cross-sectional study. Soc Sci Med. 2000 May;50(9):1317-27. doi: 10.1016/s0277-9536(99)00388-3. PMID 10728851
- [Background] Evans S, Huxley P, Gately C, Webber M, Mears A, Pajak S, Medina J, Kendall T, Katona C. Mental health, burnout and job satisfaction among mental health social workers in England and Wales. Br J Psychiatry. 2006 Jan;188:75-80. doi: 10.1192/bjp.188.1.75. PMID 16388074
- [Background] Goldstone AR, Callaghan CJ, Mackay J, Charman S, Nashef SA. Should surgeons take a break after an intraoperative death? Attitude survey and outcome evaluation. BMJ. 2004 Feb 14;328(7436):379. doi: 10.1136/bmj.37985.371343.EE. Epub 2004 Jan 20. PMID 14734519
- [Background] Karasek R, Baker D, Marxer F, Ahlbom A, Theorell T. Job decision latitude, job demands, and cardiovascular disease: a prospective study of Swedish men. Am J Public Health. 1981 Jul;71(7):694-705. doi: 10.2105/ajph.71.7.694. PMID 7246835
- [Background] Karasek R, Brisson C, Kawakami N, Houtman I, Bongers P, Amick B. The Job Content Questionnaire (JCQ): an instrument for internationally comparative assessments of psychosocial job characteristics. J Occup Health Psychol. 1998 Oct;3(4):322-55. doi: 10.1037//1076-8998.3.4.322. PMID 9805280
- [Background] McGonagle AK, Fisher GG, Barnes-Farrell JL, Grosch JW. Individual and work factors related to perceived work ability and labor force outcomes. J Appl Psychol. 2015 Mar;100(2):376-98. doi: 10.1037/a0037974. Epub 2014 Oct 13. PMID 25314364
- [Background] Siegrist J. Adverse health effects of high-effort/low-reward conditions. J Occup Health Psychol. 1996 Jan;1(1):27-41. doi: 10.1037//1076-8998.1.1.27. PMID 9547031
- [Background] Johnson JV, Hall EM. Job strain, work place social support, and cardiovascular disease: a cross-sectional study of a random sample of the Swedish working population. Am J Public Health. 1988 Oct;78(10):1336-42. doi: 10.2105/ajph.78.10.1336. PMID 3421392
- [Background] Pisanti R, van der Doef M, Maes S, Lazzari D, Bertini M. Job characteristics, organizational conditions, and distress/well-being among Italian and Dutch nurses: a cross-national comparison. Int J Nurs Stud. 2011 Jul;48(7):829-37. doi: 10.1016/j.ijnurstu.2010.12.006. Epub 2011 Jan 22. PMID 21257172
- [Background] Pomaki G, Maes S, Ter Doest L. Work conditions and employees' self-set goals: goal processes enhance prediction of psychological distress and well-being. Pers Soc Psychol Bull. 2004 Jun;30(6):685-94. doi: 10.1177/0146167204263970. PMID 15155033
- [Background] Schnall PL, Pieper C, Schwartz JE, Karasek RA, Schlussel Y, Devereux RB, Ganau A, Alderman M, Warren K, Pickering TG. The relationship between 'job strain,' workplace diastolic blood pressure, and left ventricular mass index. Results of a case-control study. JAMA. 1990 Apr 11;263(14):1929-35. PMID 2138234
- [Background] Woo M, Yap AK, Oh TG, Long FY. The relationship between stress and absenteeism. Singapore Med J. 1999 Sep;40(9):590-5. PMID 10628250
- [Background] Nielsen ML, Rugulies R, Smith-Hansen L, Christensen KB, Kristensen TS. Psychosocial work environment and registered absence from work: estimating the etiologic fraction. Am J Ind Med. 2006 Mar;49(3):187-96. doi: 10.1002/ajim.20252. PMID 16470544
- [Background] Shelledy DC, Mikles SP, May DF, Youtsey JW. Analysis of job satisfaction, burnout, and intent of respiratory care practitioners to leave the field or the job. Respir Care. 1992 Jan;37(1):46-60. PMID 10145581
- [Background] Rusli BN, Edimansyah BA, Naing L. Working conditions, self-perceived stress, anxiety, depression and quality of life: a structural equation modelling approach. BMC Public Health. 2008 Feb 6;8:48. doi: 10.1186/1471-2458-8-48. PMID 18254966
- [Background] Rosengren A, Hawken S, Ounpuu S, Sliwa K, Zubaid M, Almahmeed WA, Blackett KN, Sitthi-amorn C, Sato H, Yusuf S; INTERHEART investigators. Association of psychosocial risk factors with risk of acute myocardial infarction in 11119 cases and 13648 controls from 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):953-62. doi: 10.1016/S0140-6736(04)17019-0. PMID 15364186
- [Background] Richardson S, Shaffer JA, Falzon L, Krupka D, Davidson KW, Edmondson D. Meta-analysis of perceived stress and its association with incident coronary heart disease. Am J Cardiol. 2012 Dec 15;110(12):1711-6. doi: 10.1016/j.amjcard.2012.08.004. Epub 2012 Sep 10. PMID 22975465
- [Background] Hilton MF, Whiteford HA. Associations between psychological distress, workplace accidents, workplace failures and workplace successes. Int Arch Occup Environ Health. 2010 Dec;83(8):923-33. doi: 10.1007/s00420-010-0555-x. Epub 2010 Jul 2. PMID 20596722
- [Background] Siegrist J, Klein D, Voigt KH. Linking sociological with physiological data: the model of effort-reward imbalance at work. Acta Physiol Scand Suppl. 1997;640:112-6. PMID 9401620